CLINICAL TRIAL: NCT01661205
Title: Feasibility Trial of a Staged Epicardial & Endocardial Approach for Treatment of Patients With Persistent or Long Standing Persistent Atrial Fibrillation With Radiofrequency Ablation
Brief Title: Dual Epicardial Endocardial Persistent Atrial Fibrillation(AF) Study (Staged DEEP)
Acronym: Staged DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2012-1
Record Dates: First submitted 2012-07-11; First posted 2012-08-09 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Persistent AF; Longstanding Persistent AF; Ablation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AtriCure Bipolar System combined with a catheter ablation (Experimental): Minimally invasive procedure using the AtriCure Bipolar System plus a catheter ablation performed approximately 1-10 days apart
  Interventions: Device: Ablation procedure staged catheter ablation

INTERVENTIONS:
Device: Ablation procedure staged catheter ablation — AtriCure Bipolar System used in conjunction with a catheter ablation procedure performed 1-10 days apart

SUMMARY:
The purpose of this study is to assess the safety and technical feasibility of treating subjects with Persistent Atrial Fibrillation or Longstanding Persistent Atrial Fibrillation in a minimally invasive thoracoscopic ablation procedure utilizing the AtriCure Bipolar System, with mapping and additional lesion creation/ gap closure (as needed) provided by currently approved catheter technology, when the epicardial and endocardial phases are performed in a staged manner within 1-10 days apart, during the same hospitalization.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate how safe a less invasive cardiac surgery using the AtriCure Bipolar System in conjunction with a catheter ablation procedure performed approximately 1-10 days after, in treating atrial fibrillation, and how effective is this staged procedure. The AtriCure Bipolar System will be used to perform the less invasive cardiac surgery and a standard electrophysiology catheter, currently available, will be used to perform the catheter ablation procedure. This surgical procedure is considered less invasive because it is done through tiny surgical punctures on the sides of the chest near the ribs instead of one large surgical incision of the breast bone to completely open the chest and access the heart, and it also avoids the need for the heart-lung bypass machine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year
* Patients with symptomatic persistent or longstanding persistent AF refractory to a minimum of one Class I or III antiarrhythmic drug (AAD).
* Patients with failed catheter ablation attempts are eligible if the patients are symptomatic with persistent or longstanding persistent AF. (catheter ablation procedure must be more than 3 months prior to index procedure)
* Life expectancy of at least two years
* Patient will and able to provide informed consent
* Patient is willing and able to attend the scheduled follow-up visits

Exclusion Criteria:

* Prior Cardiothoracic Surgery
* Patient has NYHA (New York Heart Association) Class IV heart failure
* Evidence of underlying structural heart disease requiring surgical treatment
* Surgical procedure within the 30 days prior to the index procedure
* Ejection fraction < 30%
* Measured left atrial diameter > 6.0 cm
* Renal Failure
* Stroke within previous 6 months
* Known carotid artery stenosis greater than 80%
* Evidence of significant active infection or endocarditis
* Pregnant woman or women desiring to become pregnant in the next 24 months
* Presence of thrombus in the left atrium determined by echocardiography
* History of blood dyscrasia
* Contraindication to anticoagulation, based on Investigator's opinion
* Mural thrombus or tumor
* Moderate to Severe COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Stanford University Medical Center, Stanford, California
  - Colorado Springs Cardiology/Colorado Cardiac Alliance, Colorado Springs, Colorado
  - Vanderbilt Heart Institute, Nashville, Tennessee
  - Sentara Norfolk Hospital, Norfolk, Virginia
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Academic Medical Center, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject treated on September 11, 2012. A total of 31 subjects consented from 6 sites (4 USA and 2 Europe). One subject was exited from the study prior to intervention and was re-consented. Only 30 unique subjects were enrolled in the study. Twenty-six subjects treated from 5 sites.
Pre-assignment Details: Five consented subjects were withdrew prior to treatment. Three did not meet the eligibility criteria, 1 subject was withdrawn by the investigator, and 1 subject withdrew consent.
Period: Overall Study
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Started | 26
Completed | 24
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Number of Treated Subjects
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Height [Mean (Standard Deviation); unit: inches] | 71.0 (3.9)
Weight [Mean (Standard Deviation); unit: Lbs.] | 220.9 (35.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pre-specified Safety Endpoints Occurring in the First 30 Days Post-index Procedure or Hospital Discharge, Whichever is Longer.
Description: Pre-specified events include: Death; Myocardial Infarction; Stroke or TIA; Excess bleeding; Pulmonary vein stenosis; atrio-esophagael fistula; phrenic nerve paralysis; Pericardial effusion; Embolisms.
Time Frame: 30 days post-index procedure or hospital discharge
Population: Number of treated subjects. Although 26 subjects were anesthetized only 25 subjects underwent epicardial procedure per protocol. Physician decided not to treat one of the anesthetized subjects. Another case was aborted and converted to open chest cardioversion. Twenty-four patients underwent endocardial catheter procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 25
Participants | 3

2. Primary Outcome: Number of Subjects With Absence of Atrial Fibrillation
Description: Absence of atrial fibrillation (AF) at twelve month follow-up based on continuous 14 day ECG monitoring, while off all Class I and III antiarrhythmic therapy.
Time Frame: 12 month follow-up
Population: Subjects who are evaluable for primary efficacy endpoint, defined as all subjects in whom the minimally invasive staged epicardial/ endocardial ablation procedure is attempted and in whom the index-EP procedure and required post-procedure and 12 month follow-up efficacy endpoint assessment has been performed.
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 23
Participants | 18

3. Secondary Outcome: Number Subjects With Serious Device or Procedure Related Adverse Event Rate
Time Frame: 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 25
Participants
  Epicardial AF Procedure | 6
  Investigational Device | 0

4. Secondary Outcome: Number of Subjects With Acute Procedure Success
Description: Defined as subject meeting all of the following criteria upon completion of the index-EP procedure
  1. Isolation/block of all pulmonary veins (e.g. 4 of 4 veins);
  2. Bi-directional cavotricuspid isthmus block;
  3. Isolation of Box (i.e. no capture outside ablation lines connecting roof and floor lines between right-and-left pulmonary vein isolation lines);
  4. Superior Vena Cava (SVC) isolation, if encircling SVC lesion performed.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 25
Participants | 19

5. Secondary Outcome: Number of Subject Without Atrial Fibrillation
Description: AF free with or without the need of antiarrhythmic drugs
Time Frame: 6 and 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 23
Participants
  6-Months Follow-Up | 17
  12-Months Follow-Up | 19

6. Secondary Outcome: Number of Subjects With Reinterventions
Time Frame: 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 25
Participants | 8

7. Secondary Outcome: Number of Subjects With Direct Current (DC) Cardioversion
Time Frame: 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 25
Participants | 6

8. Secondary Outcome: Change in AF Based on AF Symptoms Checklist Frequency and Severity Scores
Description: Change in Atrial Fibrillation Symptom Checklist Frequency and Severity Scores. This is reported as change from Baseline.
  1. This scale has 16 items to assess frequency of occurrence on a scale: Never; Rarely; Sometimes; Often; Always. These rating correspond to numerical values of: 1, 2, 3, 4, and 5, respectively. AF Frequency range from 0 to 80 . Higher scores indicating greater symptomatology.
  2. The same items are also used to assess severity on a scale: Mild; Moderate; Severe. Corresponding to 1, 2, and 3, respectively. AF Severity score range from 0 to 48. Higher scores indicating greater symptomatology.
  3. Negative change from baseline compared to 12-months represents an improvement in AF symptomatology .
Time Frame: 12 month follow-up
Measure: Mean (Standard Deviation); unit: percentage of from baseline
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 23
percentage of from baseline
  Checklist Frequency Score | -16.3 (8.6)
  Checklist Severity Score | -12.6 (7.0)

ADVERSE EVENTS:
Time Frame: 24-months
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Serious Adverse Events (participants affected / at risk) | 12/26
Other Adverse Events (participants affected / at risk) | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System Combined With a Catheter Ablation (N=26)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Multi-organ failure (Gastrointestinal disorders) | 1 (1)
Device lead damage (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ankle operation (Surgical and medical procedures) | 1 (1)
Heart valve operation (Surgical and medical procedures) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System Combined With a Catheter Ablation (N=26)
Atrial fibrillation (Cardiac disorders) | 2 (4)
Pericardial effusion (Cardiac disorders) | 6 (6)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 2 (3)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No